CLINICAL TRIAL: NCT01519531
Title: A Randomized, Double-blind, Placebo-Controlled, Ascending Multiple-Dose Study to Evaluate the Safety, Pharmacokinetics and Pharmacodynamics of VIA-3196 in Healthy Subjects
Brief Title: Ascending Multiple-Dose Study to Evaluate VIA-3196 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Madrigal Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VIA-3196-02
Record Dates: First submitted 2012-01-24; First posted 2012-01-27 (Estimated); Last update posted 2012-12-06 (Estimated); Status verified 2012-12

CONDITIONS: Drug Safety

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- VIA-3196 (Experimental)
  Interventions: Drug: VIA-3196
- Placebo (Placebo Comparator): Multiple, ascending dosing groups (cohorts) will be evaluated.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Oral, daily-dosing for 14 days; matching number of placebo capsule(s) with active arm
  Arms: Placebo
Drug: VIA-3196 — Oral, daily dosing for 14 days
  Arms: VIA-3196

SUMMARY:
This is a single-center, randomized, double-blind, placebo-controlled, ascending multiple-dose study of VIA-3196 to evaluate the Safety, Pharmacokinetics and Pharmacodynamics of VIA-3196 in Healthy Subjects. Study dosing is organized into cohorts corresponding to escalating doses of VIA-3196 or matching placebo. Subjects will be dosed daily for 14 days.

ELIGIBILITY:
Inclusion Criteria:

* The subject must be willing and able to provide written informed consent.
* Healthy, non-smoking, males and females between the ages of 18 and 55 years of age (inclusive).
* If female, the subject is of non-child bearing potential (i.e., surgically [bilateral oophorectomy, hysterectomy, or tubal ligation] or naturally sterile [>12 consecutive months without menses]). Verify by FSH at screening as appropriate.
* Body weight > 50 kg and BMI between 18 and 30 kg/m2 (inclusive).
* LDL cholesterol ≥ 110mg/dL.

Exclusion Criteria:

* History of thyroid disorder or abnormal thyroid function tests at screening. Repeat testing is allowed once at the discretion of the Investigator. - History of unexplained syncope.
* History of hepatobiliary disease; or AST, ALT or direct bilirubin greater than the upper limit of reference range at screening.
* Positive screening test for HIV antibody, Hepatitis B surface antigen or Hepatitis C antibody.
* Abnormal screening ECG: including machine-read QTc >450 msec (confirmed by manual over read), QRS >110 msec, intermittent bundle branch block, frequent premature atrial or premature ventricular contractions, or any rhythm other than normal sinus rhythm which is interpreted by the Investigator to be clinically significant.
* History of sensitivity to a similar study drug (e.g., Karo Bio KB2115 or Metabasis MB7811), or a history of important drug or other allergy (except for untreated, asymptomatic seasonal allergies at time of dosing) unless deemed not clinically significant by the Investigator.
* History of sensitivity to thyroid medication.
* History of asthma, or intolerance to beta-blockers.
* Use of acetaminophen within 7 days before dosing and throughout the study.
* History of regular use of tobacco or nicotine containing products within the past 6 months.
* Positive urine drug screen or alcohol test at screening or Day -1.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2012-01; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events as a measure of safety and tolerability of VIA-3196 | up to 22 days
  Evaluation will start from predose (Day -1) until the follow-up visit (Day 21)

SECONDARY OUTCOMES:
Plasma concentration of VIA-3196 | 0 to 24 hours on Day 1 and Day 14
  Assessed without food
Lipid level changes following administration of VIA-3196 | Day 1 to 14

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Taub, MD, Study Director — Madrigal Pharmaceuticals
Locations (1):
- PRACS Institute (formerly Cetero Research), Fargo, North Dakota, United States